CLINICAL TRIAL: NCT01194765
Title: Distance-Based Cognitive-Behavioural Therapy for High Anxiety Sensitivity: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Janine Olthuis, Clinical Psychology PhD Candidate, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAL10-01
Record Dates: First submitted 2010-08-30; First posted 2010-09-03 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Anxiety Sensitivity
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioural Therapy (Experimental)
  Interventions: Other: Distance-based Cognitive Behavioural Therapy
- Waiting List (No Intervention)

INTERVENTIONS:
Other: Distance-based Cognitive Behavioural Therapy — Participants will engage in cognitive behavioural therapy to treat high anxiety sensitivity. Treatment will be delivered over the telephone.
  Other Names: Psychotherapy
  Arms: Cognitive Behavioural Therapy

SUMMARY:
Anxiety disorders are common pervasive conditions with serious psychosocial implications. Anxiety sensitivity (AS) is one individual characteristic that has been implicated in the onset and maintenance of anxiety disorders (Schmidt et al., 1999). AS is an enduring fear of anxiety-related arousal sensations (i.e., increased heart rate) that arises from the tendency to interpret these sensations catastrophically, believing that they will have serious physical, psychological, or social consequences (Reiss, 1991).

Research has shown the efficacy of CBT in decreasing AS among women with high AS (Watt et al., 2006). Unfortunately, access to effective psychological treatments is limited by a number of barriers such as a lack of treatment availability or qualified clinicians in an area. As such, we are conducting a randomized controlled trial (RCT) of the effectiveness of a distance-based CBT program on decreasing AS among those with high AS. A distance delivery approach (e.g., via telephone) is one way to minimize treatment barriers and increase access to care while still delivering empirically supported treatment. Recent research suggests distance delivery is promising (Lovell et al., 2006).

The RCT will consist of an eight-week structured CBT program based on Watt and Stewart's (2008) brief CBT for AS. The program will include weekly modules on psychoeducation, cognitive restructuring, interoceptive exposure, and relapse prevention. Participants with high AS will be recruited and randomly assigned to the treatment condition or wait-list control (after twelve weeks the wait-list group will receive treatment). In the treatment condition, participants will be assigned weekly reading and homework from the treatment manual. In addition, a therapist will guide them through the treatment by providing individualized support and feedback through weekly half-hour telephone sessions. Treatment outcomes will be assessed through changes in AS levels and anxiety symptoms pre- to post-treatment. Also, participants' satisfaction with the mode of treatment delivery will be assessed. We hypothesize that this treatment program will be effective in reducing high AS and anxiety symptom frequency and severity. We also expect this project to yield information about the utility of distance treatment delivery for mental health care.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* high anxiety sensitivity

Exclusion Criteria:

* cannot speak English
* illiteracy
* poor physical health (i.e., inadvisable to participate in physical exercise)
* engaged in another form of psychotherapy
* using pharmacotherapy for less than 3 months
* anyone who changes dose or type of pharmacotherapy during study
* psychosis
* suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from Pre-Treatment in Anxiety Sensitivity Level at Post-Treatment | 12 weeks
  Change from pre-treatment in participants' anxiety sensitivity level, as measured by the Anxiety Sensitivity Index - 3, will be assessed at post-treatment.

SECONDARY OUTCOMES:
Change from Pre-Treatment in Severity of Panic Symptoms at 8 Weeks | 8 weeks
  Change from pre-treatment in participants' severity of panic symptoms, as measured by sections of the Panic Attack Questionnaire - IV, will be measured at 8 weeks.
Change from Pre-Treatment in Participants' Daily Functioning at 8 Weeks | 8 weeks
  Change from pre-treatment in the amount that participants' symptoms interfere with their daily functioning, as measured by the Sheehan Disability Scale, will be assessed at 8 weeks.
Participant Satisfaction with Treatment at Post-Treatment | 12 weeks
  Participants' satisfaction with the treatment program and mode of treatment delivery will be assessed through a series of qualitative questions at post-treatment.
Change from Pre-Treatment in in General Anxiety Symptoms at 8 Weeks | 8 weeks
  Change from pre-treatment in participants' general anxiety symptoms, as measured by the Penn State Worry Questionnaire, will be assessed at 8 weeks.
Change from Pre-Treatment in Frequency of Pain-Related Anxiety Symptoms at 8 Weeks | 8 weeks
  Change from pre-treatment in participants' frequency of pain-related anxiety symptoms, as measured by the Pain Anxiety Symptom Scale - 20, will be assessed at 8 weeks.
Change from Pre-Treatment in Social Anxiety Symptoms at 8 Weeks | 8 weeks
  Change from pre-treatment in participants' level of social anxiety symptoms and amount of avoidance of social situations, as measured by the Liebowitz Social Anxiety Scale, will be assessed at 8 weeks.
Change from Pre-Treatment in Frequency and Severity of Posttraumatic Stress Symptoms at 8 weeks | 8 weeks
  For those participants who identify posttraumatic stress symptoms pre-treatment, any change in the frequency or severity of these symptoms from pre-treatment to 8 weeks will be assessed using the Modified PTSD Symptom Scale.
Change from Pre-Treatment in Drinking Motives at 8 weeks | 8 weeks
  Change from pre-treatment in participants' drinking motives (reasons for engaging in alcohol use, e.g., social, conformity, coping, or enhancement motives) at 8 weeks, as measured by the Modified Drinking Motives Questionnaire Revised, will be assessed.
Change from Pre-Treatment in Frequency of Binge Drinking at 8 weeks | 8 weeks
  Change from pre-treatment in participants' frequency of binge drinking (i.e., the number of times they imbibe 4 or more drinks within 2 hours for women or 5 or more drinks within 2 hours for men) will be assessed at 8 weeks.
Change from Pre-Treatment in Quantity and Frequency of Alcohol-Related Negative Consequences Experienced at 8 Weeks | 8 weeks
  Change from pre-treatment in the quantity and frequency of negative alcohol-related consequences experienced by participants' at 8 weeks, as measured by the Short Inventory of Problems, will be assessed.
Change from Pre-Treatment in Alcohol Expectancies at 8 Weeks | 8 weeks
  Change from pre-treatment in participants' endorsement of relief and reward alcohol expectancies, as measured by the Alcohol Craving Questionnaire, will be assessed at 8 weeks.
Change from Pre-Treatment in Anxiety Sensitivity Level at 8 weeks | 8 weeks
  Change from pre-treatment in participants' anxiety sensitivity level, as measured by the Anxiety Sensitivity Index - 3, will be assessed at 8 weeks.
Change from Pre-Treatment in Anxiety Sensitivity Level at Follow-up | 20 weeks
  Change from pre-treatment in participants' anxiety sensitivity level, as measured by the Anxiety Sensitivity Index - 3, will be assessed at follow-up.
Change from Pre-Treatment in Severity of Panic Symptoms at Post-Treatment | 12 weeks
  Change from pre-treatment in participants' severity of panic symptoms, as measured by sections of the Panic Attack Questionnaire - IV, will be measured at post-treatment.
Change from Pre-Treatment in Frequency and Intensity of Physical Exercise at Follow-up | 20 weeks
  Change from pre-treatment in participants' frequency of low-, moderate- and vigorous intensity physical exercise, as measured by the Physical Activity Measure - Modified version, will be assessed at follow-up.
Change from Pre-Treatment in in General Anxiety Symptoms at Post-Treatment | 12 weeks
  Change from pre-treatment in participants' general anxiety symptoms, as measured by the Penn State Worry Questionnaire, will be assessed at post-treatment.
Change from Pre-Treatment in in General Anxiety Symptoms at Follow-up | 20 weeks
  Change from pre-treatment in participants' general anxiety symptoms, as measured by the Penn State Worry Questionnaire, will be assessed at follow-up.
Change from Pre-Treatment in Frequency of Pain-Related Anxiety Symptoms at Post-Treatment | 12 weeks
  Change from pre-treatment in participants' frequency of pain-related anxiety symptoms, as measured by the Pain Anxiety Symptom Scale - 20, will be assessed at post-treatment.
Change from Pre-Treatment in Frequency of Pain-Related Anxiety Symptoms at Follow-up | 20 weeks
  Change from pre-treatment in participants' frequency of pain-related anxiety symptoms, as measured by the Pain Anxiety Symptom Scale - 20, will be assessed at follow-up.
Change from Pre-Treatment in Frequency of Depressive Symptoms at 8 Weeks | 8 weeks
  Change from pre-treatment in participants' frequency of depressive symptoms, as measured by the Depression Anxiety Stress Scales - 20, will be assessed at 8 weeks.
Change from Pre-Treatment in Frequency of Depressive Symptoms at Post-Treatment | 12 weeks
  Change from pre-treatment in participants' frequency of depressive symptoms, as measured by the Depression Anxiety Stress Scales - 20, will be assessed at post-treatment.
Change from Pre-Treatment in Frequency of Depressive Symptoms at Follow-up | 20 weeks
  Change from pre-treatment in participants' frequency of depressive symptoms, as measured by the Depression Anxiety Stress Scales - 20, will be assessed at follow-up.
Change from Pre-Treatment in Social Anxiety Symptoms at Post-Treatment | 12 weeks
  Change from pre-treatment in participants' level of social anxiety symptoms and amount of avoidance of social situations, as measured by the Liebowitz Social Anxiety Scale, will be assessed at post-treatment.
Change from Pre-Treatment in Social Anxiety Symptoms at Follow-up | 20 weeks
  Change from pre-treatment in participants' level of social anxiety symptoms and amount of avoidance of social situations, as measured by the Liebowitz Social Anxiety Scale, will be assessed at follow-up.
Change from Pre-Treatment in Frequency and Severity of Posttraumatic Stress Symptoms at Post-Treatment | 12 weeks
  For those participants who identify posttraumatic stress symptoms pre-treatment, any change in the frequency or severity of these symptoms from pre-treatment to post-treatment will be assessed using the Modified PTSD Symptom Scale.
Change from Pre-Treatment in Frequency and Severity of Posttraumatic Stress Symptoms at Follow-up | 20 weeks
  For those participants who identify posttraumatic stress symptoms pre-treatment, any change in the frequency or severity of these symptoms from pre-treatment to follow-up will be assessed using the Modified PTSD Symptom Scale.
Change from Pre-Treatment in Drinking Motives at Post-Treatment | 12 weeks
  Change from pre-treatment in participants' drinking motives (reasons for engaging in alcohol use, e.g., social, conformity, coping, or enhancement motives) at post-treatment, as measured by the Modified Drinking Motives Questionnaire Revised, will be assessed.
Change from Pre-Treatment in Drinking Motives at Follow-up | 20 weeks
  Change from pre-treatment in participants' drinking motives (reasons for engaging in alcohol use, e.g., social, conformity, coping, or enhancement motives) at follow-up, as measured by the Modified Drinking Motives Questionnaire Revised, will be assessed.
Change from Pre-Treatment in Frequency of Binge Drinking at Post-Treatment | 12 weeks
  Change from pre-treatment in participants' frequency of binge drinking (i.e., the number of times they imbibe 4 or more drinks within 2 hours for women or 5 or more drinks within 2 hours for men) will be assessed at post-treatment.
Change from Pre-Treatment in Frequency of Binge Drinking at Follow-up | 20 weeks
  Change from pre-treatment in participants' frequency of binge drinking (i.e., the number of times they imbibe 4 or more drinks within 2 hours for women or 5 or more drinks within 2 hours for men) will be assessed at follow-up.
Change from Pre-Treatment in Quantity and Frequency of Alcohol-Related Negative Consequences Experienced at Post-Treatment | 12 weeks
  Change from pre-treatment in the quantity and frequency of negative alcohol-related consequences experienced by participants' at post-treatment, as measured by the Short Inventory of Problems, will be assessed.
Change from Pre-Treatment in Quantity and Frequency of Alcohol-Related Negative Consequences Experienced at Follow-up | 20 weeks
  Change from pre-treatment in the quantity and frequency of negative alcohol-related consequences experienced by participants' at follow-up, as measured by the Short Inventory of Problems, will be assessed.
Change from Pre-Treatment in Alcohol Expectancies at Post-Treatment | 12 weeks
  Change from pre-treatment in participants' endorsement of relief and reward alcohol expectancies, as measured by the Alcohol Craving Questionnaire, will be assessed at post-treatment.
Change from Pre-Treatment in Alcohol Expectancies at Follow-up | 20 weeks
  Change from pre-treatment in participants' endorsement of relief and reward alcohol expectancies, as measured by the Alcohol Craving Questionnaire, will be assessed at follow-up.
Change from Pre-Treatment in Participants' Daily Functioning at Post-Treatment | 12 weeks
  Change from pre-treatment in the amount that participants' symptoms interfere with their daily functioning, as measured by the Sheehan Disability Scale, will be assessed at post-treatment.
Change from Pre-Treatment in Participants' Daily Functioning at Follow-up | 20 weeks
  Change from pre-treatment in the amount that participants' symptoms interfere with their daily functioning, as measured by the Sheehan Disability Scale, will be assessed at follow-up.
Change from Pre-Treatment in Neuroticism at Post-Treatment | 12 weeks
  Changes from pre-treatment in participants' level of neuroticism as measured by the NEO Five Factor Inventory - Neuroticism subscale
Changes from Pre-Treatment in Neuroticism at 8 weeks | 8 weeks
  Changes from pre-treatment in participants' level of neuroticsm, as measured by the NEO Five Factor Inventory - Neuroticism subscale, at 8 weeks
Change from Pre-Treatment in Neuroticism at Follow-up | 20 weeks
  Change from pre-treatment in participants' level of neuroticism, as measured by the NEO Five Factor Inventory - Neuroticism subscale, at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Janine V Olthuis, BA (Honours), Principal Investigator — Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada